CLINICAL TRIAL: NCT04781478
Title: Home Oral Care With Biorepair Implant Bioactive Gel and Chlorhexidine Gel 1% for the Improvement of Inflammatory Epidemiological Indices in Periodontal Patients: a Split-mouth Randomised Clinical Trial
Brief Title: Treatment of Periodontal Disease With Two Different Bioactive Gels for Home Oral Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-BIOCHD
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Periodontal Diseases
Keywords: split-mouth; periodontal gel; scaling and root planning; periodontal disease; dental hygiene
MeSH Terms: conditions — Periodontal Diseases | interventions — Gels

STUDY DESIGN:
Intervention Model Description: Patients are divided in two groups. Both groups are treated with non-surgical periodontal therapy (baseline and 1, 3, 6 months after the first professional oral hygiene). Patients in the first group receive Biorepair gel in quadrants Q1 and Q4 and chlorhexidine 1% gel in quadrants Q2 and Q3; for patients in the second group the situation is inverted. In this way, it is possible to compare the general periodontal condition and the quadrants treated with the two different gels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biorepair Gel (Q1-Q3) and Chlorhexidine 1% gel (Q2-Q4) (Active Comparator): The patients receive Biorepair Gel application in quadrants Q1 and Q3, whereas they receive chlorhexidine 1% gel in quadrants Q2 and Q4.
  Interventions: Other: Application of Biorepair Gel; Other: Irrigation of Chlorhexidine 1.00% gel
- Chlorhexidine 1% gel (Q1-Q3) and Biorepair Gel (Q2-Q4) (Active Comparator): The patients receive chlorhexidine 1% gel in quadrants Q1 and Q3, whereas they receive Biorepair Gel application in quadrants Q2 and Q4.
  Interventions: Other: Application of Biorepair Gel; Other: Irrigation of Chlorhexidine 1.00% gel

INTERVENTIONS:
Other: Application of Biorepair Gel — Professional application of Biorepair Gel after Scaling and Root Planing and Air-Perio polishing (glycine powders).
Other: Irrigation of Chlorhexidine 1.00% gel — Irrigation of periodontal pockets with Chlorhexidine 1.00% gel afterScaling and Root Planing and Air-Perio polishing (glycine powders).

SUMMARY:
This study is an open-label split-mouth study in which periodontal patients will be treated in order to obtain periodontal health. After non-surgical therapy and air-perio polishing, a periodontal in-situ gelling product (Biorepair Implant Bioactive gel) will be applied in periodontal pockets in two quadrants (Q1-Q3 or Q2-Q4) of the mouth of the participants. At the same time, pockets of the contralateral quadrant will be irrigated with chlorhexidine gel 1%. Patients will continue to use gels at home for the following 14 days and on the same quadrants. Professional ora hygiene session will be performed after 1, 3 and 6 months from the baseline.

Patients are divided into two groups with inverted quadrants administration in order to evaluate the improvements of periodontal inflammation indices and to assess the efficacy of Biorepair Implant Bioactive gel compared to chlorhexidine 1% gel treatment.

DETAILED DESCRIPTION:
This study is an open-label split-mouth study that aims to assess the improvement of periodontal inflammatory indices after sessions of professional oral hygiene with the administration of Biorepair Implant Bioactive Gel and Chlorhexidine gel 1%. It will also compare the efficacy of the two gel in rebalancing periodontal health.

Periodontal patients that will give the informed consent to the treatment protocol and that satisfy the eligibility criteria will undergo 4 sessions of professional oral hygiene. For each session, periodontal inflammatory indices will be recorded and professional manual and mechanical removal of supragingival and subgingival deposits of both arches will be performed, following air-perio polishing with glycine powders. At this stage, patients will be randomized and allocated to the following two groups:

* Group 1: application in periodontal pockets of quadrants Q1 and Q3 of Biorepair Implant Bioactive Gel; irrigation of periodontal pockets of quadrants Q2 and Q4 with chlorhexidine 1% gel.
* Group 2: irrigation of periodontal pockets of quadrants Q1 and Q3 with chlorhexidine 1% gel; application in periodontal pockets of quadrants Q2 and Q4 of Biorepair Implant Bioactive Gel.

Patients will continue with a home oral care protocol, using both gels for the same quadrants of their group for the following 14 days after the professional oral hygiene session.

The first session is at the baseline (T0), the second is after 1 month (T1), the third is after 3 months (T2) and the last is after 6 months (T4).

ELIGIBILITY:
Inclusion Criteria:

1. Presence of periodontal disease according to the recent 2017 classification (2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions):

   1.1 Severity from grade I onwards (grade I: clinical attachment loss of 1-2 mm, bone loss in the cervical third greater than 15%, no elements loss for periodontitis);

   1.2. Complexity from grade II onwards (grade II: maximum probing depth of 5 mm, bone loss mainly horizontally);
2. Presence of bilateral periodontal probes, both to the right and to the left of the midline incisal line.
3. Subjects who gave their written informed consent to take part of the study.

Exclusion Criteria:

* Patient with cardiac pacemaker
* Patients suffering from psychological, neurological or psychiatric disorders
* Pregnant or breastfeeding women
* Cancer patients undergoing therapy
* Patients taking bisphosphonates within the last 12 months
* Patients with low compliance or inconsistent motivation
* Drug or alcohol users
* Presence of periodontal probes exclusively on the right or left side compared to the midline incisal line

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
BOP% - Bleeding on Probing % | 1, 3 and 6 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.
PPD - Probing Pocket Depth | 1, 3 and 6 months.
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
R - Gingival recession | 1, 3 and 6 months.
  Evaluation (in mm) of the distance between the gingival margin and the amelo-cemental junction (JEC). It is the exposure of the root surface, following the apical migration of periodontal structure.
PCR% - Plaque Control Record | 1, 3 and 6 months.
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
Dental mobility (Miller, 1985) | 1, 3 and 6 months.
  It is classified using numerical values:
  0. Grade 0: oscillation within 0.2 mm; the teeth move naturally and there are no mobility problems;
  1. Grade I: horizontal mobility of the tooth from 0.2 to 1 mm;
  2. Grade II: horizontal mobility of the tooth from 1 to 2 mm;
  3. Grado III: horizontal mobility equal to or greater than 3 mm or vertical mobility of the tooth.

SECONDARY OUTCOMES:
Comparison between biorepair gel and chlorhexidine 1% gel | 1, 3 and 6 months.
  Comparing the measurements of periodontal indices in the two groups for the two different periodontal gels administered.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator